CLINICAL TRIAL: NCT04636203
Title: Burden of SARS-CoV-2 Infection in Populations With High or Low Risk of Infection
Brief Title: Burden of COVID-19 Infection in Populations With High or Low Risk of Infection
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, Professor, Neuromed IRCCS
Other Study IDs: DEP_032020
Record Dates: First submitted 2020-11-17; First posted 2020-11-19 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2 Infection; Covid19
Keywords: SARS-CoV-2; Healthcare workers; General population
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample will be taken for testing of IgM and IgG against SARS-CoV-2 and for storage in the biobank. Laboratory analyses will be performed to assess blood cell count, CRP, glucose and insulin levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General population: A sample of 3,000 men and women, residents in the territories of ASST Sette Laghi (Lombardia) and of Molise Region will be randomly selected from the municipal registries, and will be invited to participate.
- Healthcare workers (HCWs): All HCWs from the occupational registries of ASST Ospedale di Circolo Varese (Lombardia) and IRCCS Neuromed Pozzilli (Molise) will be invited to participate, up to reach 500 recruited subjects.

SUMMARY:
Introduction. Some issues remain to be elucidated about SARS-CoV-2 infection to plan prevention interventions based on scientific evidence, such as the actual prevalence of infection including subclinical and seroconverted cases, the reasons for the different spread and severity of the infection in different subjects and geographical areas as well as the impact of the COVID-19 crisis on the health of healthcare professionals and in the general population.

The aims of this project are: (i) to estimate and compare the real prevalence of the SARS-CoV-2 infection and seroconversion in two populations at high or low risk of infection,in Lombardia region and Molise region, respectively; focusing on subgroups at higher risk such as healthcare workers (HCWs); (ii) to estimate the incidence of burnout and post-traumatic stress disorder in HCWs; (iii) to identify factors associated with SARS-CoV-2 infection positivity and to follow up its mid-term effects on health.

Methods. Participants will be randomly selected from the general population of both territories and from the HCWs list of the two healthcare facilities involved. SARS-CoV-2 IgG and IgM blood levels will be measured and anamnestic data will be collected through computerized tools. Prevalence of currently or previously infected subjects and their disease status and severity will be estimated and the association with potential risk factors will be analyzed through multivariable regression analyses.

Expected results. The study will identify the burden of the infection in the general and HCWs populations. It will also identify the determinants of differences in the spread and severity of the infection, to hypothesize new preventive or therapeutic interventions. This study will provide a basis for monitoring the progress of the infection and its medium-term health consequences, Finally it will allow planning future studies, through analyses in biological samples which will be collected in dedicated biobanks.

DETAILED DESCRIPTION:
SARS-CoV-2 infection currently affects more than two million people worldwide and has caused the death of more than 150,000 people. In Lombardia there were 64.000 confirmed positive subjects (64:10,000) and 12,000 dead, with a large number of healthcare workers (HCWs) involved. However, the number of recovered is starting to rise and, thanks to the containment measures introduced, the number of new cases per day is falling. However, the situation is quite different in other part of Italy; f.i. in Molise, a southern Italy region, there is a much lower incidence of positivity and mortality: 269 confirmed positive (9:10,000) and 16 deaths.

To plan the second phase of outbreak management, waiting for the development of a vaccine and valid therapeutic tools, preventive interventions should be revisited based on evidence from the literature and from local epidemiological data. However, although the infection is now worldwide spread, some issues are still not known.

The actual number of subjects with an active or past SARS-CoV-2 infection is not known, since the approach used was based on tests performed in severe cases and in their contacts, while few investigations have been carried out on the general population. The impact of the emergency on the health of both HCWs or general population is not yet known. Furthermore, the reasons for the different spread of the infection in the North and South of the country, as well as the different characteristics of the subjects who have or have had the infection with respect to those who have not had it are not yet fully known; moreover, among the positive ones, the characteristics associated with the development of the more serious forms or the absence of symptoms, remain to be elucidated. In fact, the studies conducted so far were large studies that collected few data or were more detailed studies focused only on few hospitalized subjects.

It is therefore necessary to conduct new studies on the general population, based on large samples randomly selected from populations at high and low spread of the infection as well as in subgroups at higher risk such as HCWs, and based on a large set of collected data. The aims of this project are: (i) to estimate the real prevalence of the SARS-CoV-2 infection and seroconversion in two populations at high and low risk of infection, in a comparative way, from the territories of ASST Sette Laghi of Varese, Lombardia region (confirmed cases 18:10,000) and a region at lower prevalence of confirmed cases such as the Molise region (confirmed cases 9:10,000 subjects), also focusing on subgroups at higher risk such as healthcare workers (HCWs); (ii) to estimate the rate of burnout and post-traumatic stress disorder in HCWs during the study period; (iii) to identify factors associated with SARS-CoV-2 infection positivity and follow up at mead-term its effect on health.

Finally, the investigators will biobank biological samples for future studies, in already available specialized facilities.

(i) Cross sectional analysis in the general population Population. Residents in the territories of ASST Sette Laghi and of Molise Region will be randomly selected from the municipal registries, up to reach 3000 recruited subjects invited to participate according to protocols used in previous study.

Data collection. All people who accept the invitation at the clinics (ASST Sette Laghi Occupational Medicine in Varese, IRCCS Neuromed in Molise) will be asked to sign the informed consent and a blood sample will be taken for testing of IgM and IgG against SARS-CoV-2 and for storage in the biobank. Laboratory analyses will be performed to assess blood cell count, CRP, glucose and insulin levels.

Serum IgM and IgG antibodies will be measured with the most suitable test available at the moment of the recruitment.

To each subject an app and a website access will be given to complete questionnaires at the time of recruitment and after 6 months.

Statistical analysis. The prevalence of positivity for IgM and IgG antibodies will be calculated and the incidence during the outbreak period will be estimated. An analysis of the differences between the two geographical areas will be performed.

(ii) Cross sectional analysis on HCWs Population. All HCWs from the occupational registries of two Clinical Centers (ASST Ospedale di Circolo and IRCCS Neuromed) will be recruited.

Data collection. The HCWs who accept the invitation will be asked to sign the informed consent and a blood sample drawn for the assay of SARS-CoV-2 IgM and IgG levels and for storage in the biobank. Laboratory analyses will be performed to assess blood cell count, CRP, glucose and insulin levels, cortisol level. To each subject an app and a website access will be provided to complete questionnaires at the time of recruitment and after 6 months. In particular, they will be asked to fill: (a) Maslach Burnout Inventory (MBI), for the detection of the burnout level; (b) peritraumatic dissociative experiences questionnaire (PTEQ) and Impact of Event Scale (IES), for the detection of symptoms attributable to PTSD; (c) a reduced scale of the General Health Questionnaire (GHQ), to assess the level of psychological distress. Clinical records for SARS-CoV-2 positive participants who were hospitalized for COVID-19 will be collected in the hospital upon informed consent signature.

Statistical analysis. The prevalence of positivity to IgM and IgG antibodies will be analyzed as described in paragraph (i). Furthermore, the prevalence and incidence of MBI and PTSD disorders and the associations between the development of conditions and anamnestic, clinical and laboratory factors will be analyzed through multivariable regression analyses.

(iii) Identification of factors associated with SARS-CoV-2 infection positivity and follow up at mead-term its effect on health.

Development of a computerized application for data collection A dedicated website will be developed to allow the administration, guided by telephone aid, of specific questionnaires. Moreover, a smartphone app will be developed to follow-up participants for phase 2 COVID-19 triage and risk factors changes. Privacy and data safety will be implemented according to Italian law and guaranteed by up to date encryption standards. Questionnaire will address participants' general information (gender, age, biometrics, socio-economic status, current and previous job), lifestyles (dietary habits, smoking status, physical activity), work or leisure travel habits, previous and current diseases, pharmacological history (drugs, vaccinations and supplements), as well as specific data about COVID-19 (if they are or have been affected by the disease or they turned out to be positive to a screening). A follow up questionnaire will evaluate evolution of COVID-19 (for affected people), together with biometrics data, nutrition, physical activity, cardiovascular and neurological disorders, cognitive ability, quality of life, modifications in socio-economic level, stress, resilience.

Statistical analysis. The differences in the different variables collected between the sample of the positive subjects and a number of controls paired by sex and age, taken from the Objective 1 population will be calculated as well as the differences between the asymptomatic/paucisymptomatic non-hospitalized positives and all the other positives separated by severity (hospitalized, COVID). The analysis will be carried out through multivariate logistic regression, considering any plausibly associated variables and checking for bias from multiple tests.

ELIGIBILITY:
Inclusion Criteria:

Signing a written consent

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population Residents in the territories of ASST Sette Laghi (Lombardia) and of Molise Region will be randomly selected from the municipal registries, and will be invited to participate.
  Healthcare workers (HCWs) All HCWs from the occupational registries of ASST Ospedale di Circolo, Varese (Lombardia) and IRCCS Neuromed, Pozzilli (Molise) will be invited to partecipate
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | From December 15 2020 to June 15 2021
  To estimate and compare the real prevalence of the SARS-CoV-2 infection and seroconversion in two populations at high or low risk of infection. The knowledge of the real prevalence of currently or previously infected subjects, then the actual immunization in the general population and in HCWs, will allow to estimate the real impact of the condition and to better predict the time-course of potential new outbreaks, considering the estimated impact of the herd immunity in slowing it down
Burnout and post-traumatic stress disorder in HCWs | From December 15 2020 to June 15 2021
  To estimate the incidence of burnout and post-traumatic stress disorder in HCWs. To understand the impact of COVID-19 crisis on their health, also by quantifying their stress levels, and to set the priorities for intervention in this population subgroup (HCWs)
SARS-CoV-2 infection positivity factors/determinants | From December 15 2020 to December 15 2021
  To identify different characteristics of the subjects who have / have had the infection or the positives who have developed more serious forms will allow better understanding of the transmission pathways or the mechanism underlying the pathogenesis of the viral infection and of its manifestations, facilitating the development of new preventive or therapeutic interventions

SECONDARY OUTCOMES:
Population cohort of immunized subjects | From December 15 2020 to June 15 2022
  It is not yet known whether the immunization acquired after the infection is effective in preventing the development of the infection following a subsequent contact with the virus. This would allow to better plan the prevention interventions on the population and also to give suggestions for the research of the specific vaccine
Biobank biospecimen collection | From December 15 2020 to June 15 2022
  The biobank set up will be useful for future studies on biomarkers, which can therefore be analyzed once new hypotheses and resources are available.

CONTACTS AND LOCATIONS:
Overall Officials: Licia Iacoviello, MD, PhD, Principal Investigator — IRCCS Neuromed
Locations (2):
- Italy (2):
  - IRCCS INM Neuromed, Department of Epidemiology and Prevention, Pozzilli, IS
  - ASST Settelaghi, Varese, VA

IPD SHARING:
Plan to Share IPD: No